CLINICAL TRIAL: NCT00906581
Title: Self-guided Depression Treatment on Long-duration Spaceflights: A Continuation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); National Space Biomedical Research Institute (Other)
Responsible Party: Principal Investigator, James A. Cartreine, Instructor in Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2003P000281
Record Dates: First submitted 2009-03-19; First posted 2009-05-21 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral (Experimental): Behavioral
  Interventions: Behavioral: Computer-based Problem-Solving Treatment
- Waitlist control (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: Computer-based Problem-Solving Treatment — 6 sessions of problem-solving treatment delivered via computer
  Arms: Behavioral

SUMMARY:
Use of a computer-based treatment will reduce level of depression.

DETAILED DESCRIPTION:
Objective Depression can present a significant threat to long-duration space missions, and crews need the ability to recognize it and treat it effectively. We are developing a prototype computer-based system that includes a module for the recognition and treatment of depression. Before being used by astronauts, this system needs to be further developed and tested for efficacy in an analog population. The countermeasure we are developing is intended for use both in pre-flight training and on the International Space Station. The program has substantial Earth benefits.

Aims

1. Complete development of the module for recognizing and preventing depression. We will complete this module, moving from the prototype stage to a completed computer-based tool. We will modify the design based on data from our usability and acceptability study with astronauts at NASA Johnson Space Center. We will pilot-test the module with five participants and make revisions based on their input.
2. Develop the module for implementing computer-based Problem-Solving Treatment (PST). Currently, problem-solving treatment is done using a practitioner who guides the patient through this structured therapy and follows their progress. These practitioners are trained to administer the therapy through a formalized training program that incorporates a workbook and instructional videos. These materials are well suited for presentation via multimedia on computers to make the treatment self-guided. The PST intervention will be modified from its current video/workbook form to a computer-based form that can be used by astronauts or other professionals who are suffering from depression.
3. Evaluate the efficacy of the computer-delivered PST module for depression in a randomized, controlled trial. Hypotheses related to this aim are that, compared to a waiting-list control:

   * Individuals receiving computer-delivered PST will show a greater reduction in depression symptoms, as rated by a clinician.
   * Individuals receiving computer-delivered PST will show a greater reduction in depression, as rated by self-report.
   * A greater proportion of individuals receiving computer-delivered PST will have remitted at post-treatment.

Earth-based Applications of Research Project Depression is widespread, and effective treatments are not available to all persons who have it. This computer-based depression treatment, with simple modifications and revisions, could be adapted for use in other isolated, operational environments, such as polar research stations, submarines, commercial ships, oil rigs and underwater research facilities. Furthermore, even greater value could be derived by making similar psychosocial support systems available to the public in settings such as primary care practices, public and mental health centers, schools, social services offices, places of worship, military bases, prisons, and eventually at home or in any location, through broadband Internet.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for matching to astronaut corps population:

   * Completed 4 or more years of college or university education
   * Age 30-60
   * Has access to a personal computer and regularly uses it (at least twice per week)
2. Clinical criteria:

   * Score of 10 or higher on Hamilton Depression Inventory (which yields equivalent scores to the Hamilton Depression Rating Scale).
   * Has a diagnosis of minor depression consisting of 2 to 4 DSM-IV symptoms of depression, one of which is depressed mood or anhedonia
   * Presence of depressive symptoms for at least 2 weeks but less than 2 years
   * Patient willing to avoid or postpone the use of antidepressant drugs during the treatment portion of the study (6 weeks)

Exclusion Criteria:

1. Presence of more severe depression or dysthymia within the past 6 months (to rule out persons currently remitting from major depression)
2. Current or past diagnosis of organic mental disorder, schizophrenia, bipolar disorder, or current psychotic symptoms
3. Current suicidal ideation or any history of suicide attempt or self-injurious behavior
4. Presence of comorbid antisocial personality disorder
5. Any current substance abuse/dependence (other than nicotine or caffeine)
6. Suicidal ideation or parasuicidality
7. Current homicidal ideation
8. Recent regimen changes within the past 2 months in prescribed antidepressants, benzodiazepines, or buspirone
9. Currently receiving psychotherapy or mental health counseling
10. Exposure to PST in previous studies
11. Moderate or sever cognitive impairment (Mini Mental State Score <= 23)
12. Near terminal medical illness (physician estimates < 6 months to live)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Inventory | Pre and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: James A Cartreien, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Cartreine JA, Locke SE, Buckey JC, Sandoval L, Hegel MT. Electronic problem-solving treatment: description and pilot study of an interactive media treatment for depression. JMIR Res Protoc. 2012 Sep 25;1(2):e11. doi: 10.2196/resprot.1925. PMID 23611902